CLINICAL TRIAL: NCT07403409
Title: Effects of Scapular Repeated Contractions Facilitation Versus Hold-relax Techniques on Pain, Range of Motion and Functional Disability in Patients With Adhesive Capsulitis
Brief Title: Scapular Repeated Contractions Facilitation Versus Hold-relax Techniques in Patients With Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0196
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Adhesive Capsulitis of the Shoulder
Keywords: Adhesive Capsulitis; Scapula Repeated Contraction Facilitation Technique; scapular Hold-Relax Technique; Proprioceptive Neuromuscular Facilitation
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scapular Repeated Contraction Facilitation Technique (Experimental)
  Interventions: Other: Repeated Contraction Facilitation Technique; Other: Conventional Physical therapy Treatment for Adhesive Capsulitis
- Scapular Hold-Relax Technique (Active Comparator)
  Interventions: Other: Hold-Relax Technique; Other: Conventional Physical therapy Treatment for Adhesive Capsulitis

INTERVENTIONS:
Other: Repeated Contraction Facilitation Technique — Repeated contraction facilitation on scapula in two diagonal patterns (D1&D2) were performed .D1 consisted of anterior elevation and posterior depression and D2 consisted of posterior elevation and anterior depression. Isotonic contraction of muscles against the resistance throughout the active ROM was performed.3 sets of 10 repetitions were performed with 20 seconds of rest interval.
  Arms: Scapular Repeated Contraction Facilitation Technique
Other: Hold-Relax Technique — Hold -Relax on scapula in two diagonal patterns (D1&D2) were performed .D1 consisted of anterior elevation and posterior depression and D2 consisted of posterior elevation and anterior depression in which restricted muscles were contracted isometrically with 5 sec hold followed by relaxation into new range .3 sets of 10 repetitions were performed with 20 seconds of rest interval.
  Arms: Scapular Hold-Relax Technique
Other: Conventional Physical therapy Treatment for Adhesive Capsulitis — Moist heat pack for 15-20 mins Therapeutic Ultrasound at 1MHz for 8-10 mins in continuous mode with the intensity of 1.5W/cm2 Active Assisted Shoulder for abduction, flexion, internal rotation and external rotation with 3 sets of 15 repetitions 4days/week for 4 weeks Wall slides, Finger ladder exercises, Wand exercises and home exercises were performed.3x15 repetitions with 2 min rest interval for 4 sessions per week for four weeks for each exercise Maitland Glenohumeral Joint Mobilization with 2-3 oscillations per second for 30 seconds for 5 sets 4 times a week in caudal and posteroanterior direction was applied for 4 weeks.

SUMMARY:
The study was conducted to determine the effects of scapular repeated contractions facilitation versus hold-relax techniques on pain, range of motion and functional disability in patients with adhesive capsulitis

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed stage 2 of Adhesive Capsulitis (>4-12 months)
* Difficulties in 2 or more movements: external rotation, abduction, flexion or internal rotation presenting limitation of more than 30 degrees
* Patients having diagnosed Diabetes Mellitus type 2
* Capsular pattern of restriction
* Unilateral involvement of the shoulder
* Patients who are not taking any pain killer

Exclusion Criteria:

* Surgical history of affected shoulder
* History of trauma or fracture in affected shoulder
* Cervical neuropathy or any other disorders of cervical spine, elbow and wrist
* Any Neurological disorders such as stroke or parkinsonism
* Any systemic disease such as rheumatoid arthritis, osteoporosis and malignancies in shoulder region
* Intra-articular injection
* Open wound or skin infection
* Manipulation under anesthesia
* Recurrent dislocation or subluxation
* Shoulder injuries such as rotator cuff tear, or tendon calcification

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2025-01-18 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | At base line and end of 4 weeks
  Patient level of pain was assessed using this scale. This scale ranges from 0 to 10. 0 indicates "no pain" ,1- 3 indicates mild pain ,4-6 indicates moderate pain and 7-10 indicates "worst pain". NPRS have shown high test-retest reliability (r = 0.96 and 0.95, respectively) MCID value of NPRS is 2-3
Shoulder Pain And Disability Index | from baseline to end of 4 weeks
  SPADI was used to assess functional disability. It has 13 items, with 5 items for pain and 8 items for disability

SECONDARY OUTCOMES:
ROM shoulder flexion | 4th week
  changes from baseline ROM of shoulder flexion was taken
ROM shoulder abduction | 4th week
  changes from baseline ROM of shoulder was taken
ROM shoulder external rotation | 4th week
  changes from baseline ROM of shoulder external rotation was taken
ROM shoulder internal rotation | 4th week
  changes from baseline ROM of shoulder internal rotation was taken

CONTACTS AND LOCATIONS:
Overall Officials: Ameena Amjad, Ph.D, Principal Investigator — Riphah International University
Locations (1):
- Rasool Medical Complex Gujrat, Dhok Gujra, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joshi D, Chitra J. Effect of scapular proprioceptive neuromuscular facilitation on shoulder pain, range of motion, and upper extremity function in hemiplegic patients: A randomized controlled trial. Indian Journal of Health Sciences and Biomedical Research KLEU. 2017;10(3):276-82.
- [Background] Chitra J, Joshi D. Effect of scapular hold-relax technique on shoulder pain in hemiplegic subjects: A randomized controlled trial. Physiotherapy-The Journal of Indian Association of Physiotherapists. 2017;11(2):49-52.
- [Background] Mishra N, Mishra A, Charaniya P. Effect of scapular proprioceptive neuromuscular facilitation on pain and disability in patients with adhesive capsulitis. Int J Yogic Hum Mov Sports Sciences. 2019;4(1):995-1000.
- [Background] Saeed M, Hafeez S, Asad F, Haider W, Nawaz S, Kocub S. Comparison of scapular proprioceptive neuromuscular facilitation and myofascial release techniques on pain and function in scapular dyskinesia associated with adhesive capsulitis: Scapular dyskinesia associated with adhesive capsulitis. Pakistan BioMedical Journal. 2022:123-7.
- [Background] Bhavika PG, Vinosh Kumar P. Effect of Scapular Proprioceptive Neuromuscular Facilitation versus Scapular Mobilization on Pain and function in adhesive capsulitis-A Pragmatic Randomized Clinical Trial. INTI JOURNAL. 2023;2023(64):1-6.
- [Background] Akgüller T, Akbaba YA, Taşkıran H. The effect of scapular proprioceptive neuromuscular facilitation techniques on pain and functionality in patients with subacromial impingement syndrome: a randomized controlled trial. Physikalische Medizin, Rehabilitationsmedizin, Kurortmedizin. 2023;33(03):149-61.
- [Background] Shaikh SB, Ganvir SS. Effect of 4 Weeks of Scapular Proprioceptive Neuromuscular Facilitation on Scapular Alignment and Upper Extremity Motor Performance in Patients with Stroke: A Repeated Measure Design. Medical Journal of Dr DY Patil Vidyapeeth. 2023;16(Suppl 2):S228-S34.
- [Background] Ragapriyaa R, Kamalakannan M, Anitha A, Ramana K. Effect of Scapular Clock Exercise Versus Scapular PNF Exercise on Pain and ROM for Anterior Capsular Stiffness of Shoulder Joint. Indian Journal of Physiotherapy & Occupational Therapy. 2024;18.
- [Background] Cellatoğlu H, Kaygısız BB. Effect of proprioceptive neuromuscular facilitation (PNF) technique on posture, balance and gait characteristics of older adults with scapular dyskinesis: a randomized controlled trial. PeerJ. 2025;13:e19718.
- [Background] Butt MS, Tanveer F. Effects of scapular proprioceptive neuromuscular facilitation techniques in addition to routine physical therapy on clinical outcomes in patients with adhesive capsulitis: A randomized controlled trial. The Healer Journal of Physiotherapy and Rehabilitation Sciences. 2022;2(1):78-87.
- [Background] Ghias S, Saeed H, Ahmed M, Faisal M, Solangi TA, Asim HAB, et al. Effectiveness of PNF Pattern in Regular Physical Therapy Sessions on Functional Mobility in Frozen Shoulder: PNF Pattern in Frozen Shoulder Therapy. THE THERAPIST (Journal of Therapies & Rehabilitation Sciences). 2024:46-50.
- [Background] Lin P, Yang M, Huang D, Lin H, Wang J, Zhong C, et al. Effect of proprioceptive neuromuscular facilitation technique on the treatment of frozen shoulder: a pilot randomized controlled trial. BMC musculoskeletal disorders. 2022;23(1):367
- [Background] Zhang EJX, Lam YX, Lim WSR, Lie DTT. Effect of proprioceptive neuromuscular facilitation on efficacy and pain relief for symptomatic shoulder conditions: a meta-analysis. Journal of Orthopaedic Reports. 2025;4(1):100541.